CLINICAL TRIAL: NCT01665287
Title: Cerebral Oximetry in Newborns - Comparing INVOS 5100 and FORE-SIGHT Cerebral Oximeters Absolute Values, Sensitivity for Low Oxygen Levels and Reproducibility..
Brief Title: Cerebral Oximetry in Newborns - Comparing INVOS 5100 and FORE-SIGHT Cerebral Oximeters
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: The Augustinus Foundation, Denmark. (Other)
Responsible Party: Principal Investigator, Gorm Greisen, Professor, MD, Rigshospitalet, Denmark
Other Study IDs: 300712FORVOS
Record Dates: First submitted 2012-08-13; First posted 2012-08-15 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2013-01

CONDITIONS: Near Infrared Spectroscopy
Keywords: Cerebral Oximetry; Near infrared spectroscopy; Fullterm; Infant

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Regional tissue oxygenation (rStO2) can be monitored by near infrared spectroscopy. The commercial devices FORE-SIGHT (CASMED) and INVOS (COVIDIEN) will be used simultaneously to test for their relative sensitivity for low oxygen levels just after birth on term infants born by elective cesarean section. Reproducibility will be examined by replacements of the sensors six times the next day when the infant is stable and quiet. Neonatal sensors will be used.

ELIGIBILITY:
Inclusion Criteria:

* Term infants (age more than 37 weeks of gestation)
* Elective cesarean section after an uncomplicated pregnancy

Exclusion criteria:

* Thick hair that makes good measurements difficult/impossible
* Obvious malformations or syndrome
* Complications in relation to the cesarean section
* Depression after birth (APGAR < 8 after 1 minute)

Max Age: 2 Minutes | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Term infants born by elective cesarian section.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2012-08; Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Cerebral oxygenation | 10 minutes
  The sensors of both instruments will be placed on each side of the head. They will be held by hand or by self-adhesive tape as appropriate.
  Curve fitting will be used to describe the rapid increase of oxygenation after birth. Estimated cerebral oxygenation at 3 min (hypoxia) and 10 min (normoxia) will be used to compare the two instruments.

SECONDARY OUTCOMES:
Reproducibility | 10 minutes
  The sensor will be placed 6 times alternating on each frontoparietal region and held by hand, obtaining 30 seconds of signal for each placement. The placements will be in the same region but not in exactly the same spot. This will be done for both devices.

CONTACTS AND LOCATIONS:
Overall Officials: Gorm Greisen, Professor, Principal Investigator — Not relevant
Locations (1):
- Department of Neonatology, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Background] Noori S, Wlodaver A, Gottipati V, McCoy M, Schultz D, Escobedo M. Transitional changes in cardiac and cerebral hemodynamics in term neonates at birth. J Pediatr. 2012 Jun;160(6):943-8. doi: 10.1016/j.jpeds.2011.12.008. Epub 2012 Jan 11. PMID 22244465
- [Background] Kratky E, Pichler G, Rehak T, Avian A, Pocivalnik M, Muller W, Urlesberger B. Regional cerebral oxygen saturation in newborn infants in the first 15 min of life after vaginal delivery. Physiol Meas. 2012 Jan;33(1):95-102. doi: 10.1088/0967-3334/33/1/95. PMID 22173332
- [Background] Urlesberger B, Kratky E, Rehak T, Pocivalnik M, Avian A, Czihak J, Muller W, Pichler G. Regional oxygen saturation of the brain during birth transition of term infants: comparison between elective cesarean and vaginal deliveries. J Pediatr. 2011 Sep;159(3):404-8. doi: 10.1016/j.jpeds.2011.02.030. Epub 2011 Apr 9. PMID 21481417
- [Background] Urlesberger B, Grossauer K, Pocivalnik M, Avian A, Muller W, Pichler G. Regional oxygen saturation of the brain and peripheral tissue during birth transition of term infants. J Pediatr. 2010 Nov;157(5):740-4. doi: 10.1016/j.jpeds.2010.05.013. Epub 2010 Jun 17. PMID 20955848